CLINICAL TRIAL: NCT05267015
Title: PRF for Treating Maxillary Gingival Recessions: A Split-mouth, Randomized, Controlled Clinical Trial
Brief Title: PRF for Treating Maxillary Gingival Recession
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arab American University (Palestine) (Other)
Responsible Party: Principal Investigator, Mahmoud Abu-Ta'a, Associate Professor, Arab American University (Palestine)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ArabAmericanU
Record Dates: First submitted 2022-02-14; First posted 2022-03-04 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-02

CONDITIONS: Gingival Recession
Keywords: connective tissue graft; PRF membrane; gingival recession
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- coronally advanced flap with connective tissue graft (Active Comparator): After randomization a subepithelial connective tissue graft along with coronally advanced flap is applied to one maxillary quadrant to cover the recession.
  Interventions: Procedure: Gingival coverage using coronally advanced flap and a connective tissue graft
- coronally advanced flap with platelet rich fibrin membranes (Experimental): After randomization platelet rich fibrin membranes along with coronally advanced flap are applied to the other maxillary quadrant to cover the recession.
  Interventions: Procedure: Gingival coverage using coronally advanced flap and platelet rich fibrin membranes

INTERVENTIONS:
Procedure: Gingival coverage using coronally advanced flap and a connective tissue graft — A coronally advanced flap is applied for recession coverage in the maxilla in a split-mouth randomized trial using a subepithelial connective tissue graft
  Arms: coronally advanced flap with connective tissue graft
Procedure: Gingival coverage using coronally advanced flap and platelet rich fibrin membranes — A coronally advanced flap is applied for recession coverage in the maxilla in a split-mouth randomized trial using platelet rich fibrin membranes
  Arms: coronally advanced flap with platelet rich fibrin membranes

SUMMARY:
This is a split-mouth, randomized, controlled clinical trial that aims to evaluate the clinical efficacy of platelet-rich fibrin (PRF) membranes in conjunction with coronally advanced flap (CAF) in treating maxillary gingival recession defects.

ELIGIBILITY:
Inclusion Criteria:

* Greater than 18 years old
* Bilateral Miller class I + II recession in the upper jaw

Exclusion Criteria:

* Smokers
* Patients with systemic diseases that could interfere with the healing
* Patients undergoing bisphosphonate therap .Patients who previously received radiation therapy of the jaws.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-01-03 (Actual); Primary Completion 2021-08-15 (Actual); Study Completion 2021-11-14 (Actual)

PRIMARY OUTCOMES:
Increase in gingival height (recession coverage) | six weeks
  The measurements of the increase in gingival height (recession coverage) using a linear evaluation (corono-apical direction) with a periodontal probe (Merrit-B; Hu-Friedy, Chicago, IL, USA) at the interventions sites to the nearest 0.5 mm. Registration of the recession height was done before treatment and after 6 weeks.
Shrinkage in gingival height | six months
  To assess the shrinkage of the gingival height, the amount of gingival height vestibular to the treated teeth in a corono-apical direction was measured after the surgery and after six months.

SECONDARY OUTCOMES:
Postoperative pain visual analog scores (VAS) and surgery time | two weeks
  This questionnaire used 100 mm visual analog scores VAS to evaluate the amount of pain, ranging from 0 (no pain) to 10 (worst pain imaginable), and the amount of swelling. Patients were asked to fill in the VAS scales at day 7 and day 14 at suture removal. The time of surgery was measured of both treatment options. Timing started at the moment of first incision until the last suture.

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud F Abu-Ta'a, Periodontist, Principal Investigator — Head of Department
Locations (1):
- Arab American University, Ramallah, Palestinian Territories

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abu-Ta'a M. Advanced Platelet-Rich Fibrin and Connective Tissue Graft for Treating Marginal Tissue Recessions: A Randomized, Controlled Split-Mouth Study. Cureus. 2023 Mar 4;15(3):e35761. doi: 10.7759/cureus.35761. eCollection 2023 Mar. PMID 36879584